CLINICAL TRIAL: NCT00016354
Title: Phase I Study of Continuous Weekly Dosing of Dimethyl Benzoylphenylurea (BPU) in Patients With Solid Tumors Not Responding to Conventional Therapy
Brief Title: Benzoylphenylurea in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0072 CDR0000068625; U01CA070095 (NIH); P30CA006973 (NIH); JHOC-J0072 (Other: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins); NCI-1351 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- benzoylphenylurea (Experimental)
  Interventions: Drug: benzoylphenylurea

INTERVENTIONS:
Drug: benzoylphenylurea

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of benzoylphenylurea in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of benzoylphenylurea in patients with advanced solid tumors.
* Evaluate the acute and chronic toxicity profile of this regimen in these patients.
* Evaluate the pharmacokinetics and metabolites of this regimen and any potential correlation with pharmacodynamic effects in these patients.
* Determine the antitumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral benzoylphenylurea (BPU) once weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BPU until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience a dose-limiting toxicity. Once the MTD is determined, 12 additional patients are accrued and treated with BPU as above to confirm the MTD.

Patients are followed for 30 days.

PROJECTED ACCRUAL: Approximately 18-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy

  * Metastatic or unresectable
  * No effective standard curative or palliative measures exist
* No known CNS or brain metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* SGOT/SGPT normal

Renal:

* Creatinine normal
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No uncontrolled ventricular arrhythmia
* No myocardial infarction within the past 3 months
* No superior vena cava syndrome

Neurologic:

* No grade 1 or greater peripheral neuropathy
* No uncontrolled major seizure disorder
* No spinal cord compression

Other:

* No active serious infection requiring IV antibiotics
* No concurrent uncontrolled illness
* No concurrent unstable or serious medical condition
* No chronic diarrhea or malabsorption
* No history of allergic reactions to compounds similar in chemical or biological composition to benzoylphenylurea
* No psychiatric illness or social situation that would preclude study compliance
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy
* No concurrent growth factors during first 2 courses of study
* Concurrent epoetin alfa allowed

Chemotherapy:

* At least 28 days since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy

Radiotherapy:

* At least 28 days since prior large-field radiotherapy
* Prior palliative radiotherapy for painful bone metastases allowed
* No concurrent radiotherapy, including palliative or whole-brain radiotherapy for CNS disease

Surgery:

* At least 28 days since prior major surgery

Other:

* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial agents or therapies for the malignancy
* No other concurrent investigational agents
* Concurrent bisphosphonates allowed if bone metastases are not only site of measurable or evaluable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2001-03; Primary Completion 2004-08 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio C. Wolff, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Messersmith WA, Rudek MA, Baker SD, Zhao M, Collins C, Colevas AD, Donehower RC, Carducci MA, Wolff AC. Phase I study of continuous weekly dosing of dimethylamino benzoylphenylurea (BPU) in patients with solid tumours. Eur J Cancer. 2007 Jan;43(1):78-86. doi: 10.1016/j.ejca.2006.09.006. Epub 2006 Nov 3. PMID 17084620
- [Result] Messersmith WA, Baker SD, Donehower RC, et al.: Phase I study of continuous weekly dosing of dimethyl benzoylphenylurea (BPU) in patients with solid tumors. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-815, 2003.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nineteen patients were enrolled between August 2001 and July 2004 at Johns Hopkins.
Pre-assignment Details: Patients were excluded if they had known brain metastases, active infections, chronic diarrhoea, malabsorption, peripheral neuropathy >grade 1 (NCI CTC v2), pregnancy, HIV infection, or serious concurrent medical conditions.
Groups:
- Benzoylphenylurea 5 mg: Benzoylphenylurea dose level of 5 mg; Dose level 1
- Benzoylphenylurea 10 mg: Benzoylphenylurea dose level of 10 mg; Dose level 2
- Benzoylphenylurea 20 mg: Benzoylphenylurea dose level of 20 mg; Dose level 3
- Benzoylphenylurea 40 mg: Benzoylphenylurea dose level of 40 mg; Dose level 4
- Benzoylphenylurea 80 mg: Benzoylphenylurea dose level of 80 mg; Dose level 5
- Benzoylphenylurea 160 mg: Benzoylphenylurea dose level of 160 mg; Dose level 6
- Benzoylphenylurea 320 mg: Benzoylphenylurea dose level of 320 mg; Dose level 7
- Benzoylphenylurea Dose Level of 150 mg: Benzoylphenylurea dose level of 150 mg; Dose level 8 (for this dose level, a 25 mg capsule was used. At all previous dose levels, a 5 mg capsule was administered.)
Period: Overall Study
Arm/Group | Benzoylphenylurea 5 mg | Benzoylphenylurea 10 mg | Benzoylphenylurea 20 mg | Benzoylphenylurea 40 mg | Benzoylphenylurea 80 mg | Benzoylphenylurea 160 mg | Benzoylphenylurea 320 mg | Benzoylphenylurea Dose Level of 150 mg
Started | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 7
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Benzoylphenylurea: BPU, administered over a dose range of 5-320 mg
Arm/Group | Benzoylphenylurea
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Determine Maximum Tolerated Dose of BPU
Description: Toxicity was assessed weekly during the first 2 cycles, and monthly thereafter, using the National Cancer Institute Common Toxicity Criteria (NCI CTCv2). Dose limiting toxicity (DLT) was defined as dose delays >2 weeks, grade 4 haematologic toxicity (except grade 4 neutropenia lasting <5 days), or grade 3 nonhaematologic toxicity. The maximum tolerated dose (MTD) is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience a dose-limiting toxicity.
Time Frame: 4 weeks (1 course of treatment for each subject)
Population: Participants that completed at least 1 cycle of BPU.
Measure: Number; unit: milligrams (mg)
Arm/Group | Benzoylphenylurea
Number analyzed (Participants) | 19
milligrams (mg) | 150

2. Secondary Outcome: Number of Patients With Adverse Events
Time Frame: every 4 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of BPU
Time Frame: 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Test for Antitumor Activity in Blood and Tissue
Time Frame: baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: every 4 weeks
Description: Toxicity was assessed weekly during the first 2 cycles, and monthly thereafter, using the NCI CTCv2.
Arm/Group | Benzoylphenylurea
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benzoylphenylurea (N=19)
Neutropenic fever (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benzoylphenylurea (N=19)
Anemia (Hemoglobin) (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Platelets) (Blood and lymphatic system disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Headache (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes